CLINICAL TRIAL: NCT02991261
Title: A Randomized, Open-Label, Single-Dose Bioavailability Study of SPARC001in Healthy, Adult Volunteers Under Fed and Fasted Conditions"
Brief Title: Bioavailability Study of SPARC001 (Study 2) in Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sun Pharma Advanced Research Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CLR_16_29
Record Dates: First submitted 2016-12-08; First posted 2016-12-13 (Estimated); Last update posted 2019-05-03 (Actual); Status verified 2019-05

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- SPARC001 type I (Experimental): Treatment type I
  Interventions: Drug: SPARC001 type I; Drug: SPARC001 type II; Drug: Reference001 type I; Drug: Reference001 type II
- SPARC001 type II (Experimental): Treatment type II
  Interventions: Drug: SPARC001 type I; Drug: SPARC001 type II; Drug: Reference001 type I; Drug: Reference001 type II
- Reference001 type I (Active Comparator): Hydrocodone-Acetaminophen
  Interventions: Drug: SPARC001 type I; Drug: SPARC001 type II; Drug: Reference001 type I; Drug: Reference001 type II
- Reference type II (Active Comparator): Hydrocodone-Acetaminophen
  Interventions: Drug: SPARC001 type I; Drug: SPARC001 type II; Drug: Reference001 type I; Drug: Reference001 type II

INTERVENTIONS:
Drug: SPARC001 type I — Treatment type I
Drug: SPARC001 type II — Treatment type II
Drug: Reference001 type I — Hydrocodone-acetaminophen
Drug: Reference001 type II — Hydrocodone Acetaminophen

SUMMARY:
The objective of the study is to determine the relative bioavailability, safety and tolerability of SPARC001 and Reference001 in healthy, adult, male and female subjects

ELIGIBILITY:
Inclusion Criteria:

1. Adult, male and female volunteers, 18 to 55 years of age, inclusive, at first Check-In Visit
2. Body mass index (BMI) ≥18 to ≤30 kg/m2 and total body weight >50 kg (110 lbs) at Screening
3. All female subjects must have a negative serum pregnancy test at Screening and at each Check-in Visit
4. Medically healthy on the basis of medical history and physical examination (including but not limited to an evaluation of the cardiovascular, gastrointestinal, respiratory and central nervous systems), as determined by the Investigator at Screening and each Check-In Visit.

Exclusion Criteria:

1. Females who are pregnant, lactating, or likely to become pregnant during the study
2. Life-time history and/or recent evidence of alcohol or drug/substance abuse disorder
3. Subjects who need to maintain mental alertness throughout the study
4. Subjects determined by the investigator to have any medical condition that could jeopardize their health or prejudice the results

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2017-02-06 (Actual); Primary Completion 2017-03-15 (Actual); Study Completion 2017-04-01 (Actual)

PRIMARY OUTCOMES:
AUC | 48 hours
Cmax | 48 hours

SECONDARY OUTCOMES:
Adverse event | 25 days

CONTACTS AND LOCATIONS:
Locations (1):
- SPARC Site 01, Secaucus, New Jersey, United States